CLINICAL TRIAL: NCT07109258
Title: Effect of Dexamethasone on Labour Induction in Term Pregnancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelfatah Mohamed Kamel Eldesouky, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS-552-2024
Record Dates: First submitted 2025-07-07; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Labor Induction
Keywords: Labor Induction; Dexamethasone; Misoprostol; Term pregnancies
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Injections, Intramuscular; Misoprostol

STUDY DESIGN:
Intervention Model Description: 1. Group A: They will receive one dose of IM dexamethasone sodium phosphate 8 mg (2 mL).
  2. Group B: They will receive vaginal misoprostol 25 μg tablets every 6 h, up to 4 tablets, for a maximum duration of 24 h.
  3. Group C: They will receive one dose of IM dexamethasone sodium phosphate 8mg (2mL) with the first dose of vaginal misoprostol 25 μg tablets that will be given every 6 h, up to 4 tablets, for a maximum duration of 24 h.
     * Regarding group A,B and C we will wait 24hrs after the last dose, then reassessment by senior obstetrician will be done and if induction is unsuccessful it'll be determined whether the patient is for either CS or second 24hr attempt at induction by misoprostol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): They will receive one dose of IM dexamethasone sodium phosphate 8 mg (2 mL).
  Interventions: Drug: Dexamethasone (Decadron) 8mg IM injection
- Group B (Active Comparator): They will receive vaginal misoprostol 25 μg tablets every 6 h, up to 4 tablets, for a maximum duration of 24 h.
  Interventions: Drug: Misoprostol 25 mcg
- Group C (Experimental): They will receive one dose of IM dexamethasone sodium phosphate 8mg (2mL) with the first dose of vaginal misoprostol 25 μg tablets that will be given every 6 h, up to 4 tablets, for a maximum duration of 24 h.
  Interventions: Drug: Both Misoprostol 25 mcg & Dexamethasone 8mg IM injection

INTERVENTIONS:
Drug: Dexamethasone (Decadron) 8mg IM injection — one dose of IM dexamethasone sodium phosphate 8 mg (2 mL) given at the start of labour induction
  Arms: Group A
Drug: Misoprostol 25 mcg — vaginal misoprostol 25 μg tablets every 6 h, up to 4 tablets, for a maximum duration of 24 h.
  Arms: Group B
Drug: Both Misoprostol 25 mcg & Dexamethasone 8mg IM injection — one dose of IM dexamethasone sodium phosphate 8mg (2mL) with the first dose of vaginal misoprostol 25 μg tablets that will be given every 6 h, up to 4 tablets, for a maximum duration of 24 h.
  Arms: Group C

SUMMARY:
The aim of the study is to assess the effect of dexamethasone on labour induction in term pregnancies.

Primary outcome:

The interval between initiation of induction and beginning of the active phase of labour.

Secondary outcomes:

* Duration of active phase of labour (starting with cervical dilatation of 4-5 cm up to full cervical dilatation).
* Duration of second stage of labour
* Mode of delivery.
* Fetal outcome.

Group A:

Will receive one dose of IM dexamethasone sodium phosphate 8 mg (2 mL).

Group B:

Will receive vaginal misoprostol 25 μg tablets every 6 h, up to 4 tablets, for a maximum duration of 24 h.

Group C:

Will receive one dose of IM dexamethasone sodium phosphate 8mg (2mL) with the first dose of vaginal misoprostol 25 μg tablets that will be given every 6 h, up to 4 tablets, for a maximum duration of 24 h.

DETAILED DESCRIPTION:
* Study type: Randomized Controlled Trial
* Population of study:

Pregnant women above 18 years of age, eligible for induction of labour.

● Study location: Cairo University Obstetrics & Gynecology Hospital (Kasr Al-Ainy)

* Methodology in details:

  * Every subject will be subjected to:
  * Written consent.
  * Complete history to exclude systemic disorders, congenital fetal malformation and contraindications for vaginal delivery.
  * General examination of the patients including pulse, blood pressure and body mass index, [weight (kg)/ height (m2)] (20-25) normal weight, (25-30) overweight, (30-35) obese, (35-40) very obese and >40 morbid obese.
  * Abdominal examination including presentation, station of fetal head, fetal heart rate, uterine contractions and exclusion of multiple pregnancies.
  * Local examination to determine cervical dilatation at the beginning of intervention, presenting part, station of fetal head, pelvic adequacy and Bishop scoring.
  * Sonographic examination including assessment of fetal well-being by biophysical profile.
  * Patients will be randomly assigned to three groups using simple randomization via computer-generated random numbers will be used.
  * The women will be divided into three groups:

    1. Group A: They will receive one dose of IM dexamethasone sodium phosphate 8 mg (2 mL).
    2. Group B: They will receive vaginal misoprostol 25 μg tablets every 6 h, up to 4 tablets, for a maximum duration of 24 h.
    3. Group C: They will receive one dose of IM dexamethasone sodium phosphate 8mg (2mL) with the first dose of vaginal misoprostol 25 μg tablets that will be given every 6 h, up to 4 tablets, for a maximum duration of 24 h.
* Regarding group A,B and C the investigators will wait 24hrs after the last dose, then reassessment by senior obstetrician will be done and if induction is unsuccessful it'll be determined whether the patient is for either CS or second 24hr attempt at induction by misoprostol.
* Primary outcome:

The interval between initiation of induction and beginning of the active phase of labour.

* Secondary outcomes:

  * Duration of active phase of labour (starting with cervical dilatation of 4-5 cm up to full cervical dilatation).
  * Duration of second stage of labour
  * Mode of delivery.
  * Fetal outcome.
* Sample size Assuming that the mean interval between the start of induction and the beginning of the active phase among cases 2.87±1.57 hours versus 3.8±1.72 hours among controls, so a minimum sample of 150 patients, divided into three equal groups (50 patients each), will achieve 80% power at 0.05 significance level. Sample size calculated using OpenEpi, Version 3, open source calculator-(SSMean).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Nulliparous.
* Vertex presentation.
* Singleton pregnancy.
* Gestational age ≥ 39 weeks according to a reliable date for the last menstrual period or a first-trimester ultrasound evaluation.
* No contraindication for vaginal delivery.

Exclusion Criteria:

* Indication for cesarean section e. g. Placenta previa, intrauterine growth retardation, non-vertex presentation and previous cesarean section.
* Maternal medical disorders as diabetes mellitus and severe pre-eclampsia.
* Preterm labour and preterm rupture of membranes.
* Gestational age <39 weeks of gestation.
* Fetal macrosomia > 4kg (estimated by u/s).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The interval between initiation of induction and beginning of the active phase of labour. | The interval between initiation of induction and beginning of the active phase of labour, assessed hourly up to 24 hours.
  Assessed hourly

SECONDARY OUTCOMES:
Duration of active phase of labour (starting with cervical dilatation of 4-5 cm up to full cervical dilatation). | Duration of active phase of labour (starting with cervical dilatation of 4-5 cm up to full cervical dilatation), assessed hourly up to 24 hours.
  Assessed hourly
Duration of second stage of labour | Recorded immediately with delivery of the baby
Mode of delivery | After induction attempt (24 hours)
  Vaginal or Cesarean
Fetal outcome | At 1 and 5 minutes after delivery
  APGAR score
Fetal Outcome | Recorded within 24 hours after delivery
  NICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospital (Kasr Al Ainy), Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Confidentiality

REFERENCES:
- [Background] Vilas-Boas LS, Sanches MPR, Araujo Junior E, Peixoto AB, Mattar R, Santos LRRD, Pares DBDS, Sun SY. Evaluation of the efficacy of labor induction with vaginal misoprostol in a low-risk pregnant women population. Rev Assoc Med Bras (1992). 2024 Jul 19;70(7):e20240132. doi: 10.1590/1806-9282.20240132. eCollection 2024. PMID 39045936
- [Background] Laloha F, Asiabar NM, Barikani A, Movahed F, Haj Seyed Javadi E. Effect of Intravenous Dexamethasone on Preparing the Cervix and Labor Induction. Acta Med Iran. 2015;53(9):568-72. PMID 26553085
- [Background] Mohaghegh Z, Faal Siahkal S, Bahmaei H, Sharifipour F, Leyli EK, Zahedian M. The effect of dexamethasone on labor induction: a systematic review. BMC Pregnancy Childbirth. 2021 Aug 17;21(1):563. doi: 10.1186/s12884-021-04010-1. PMID 34404372
- [Background] Kavanagh J, Kelly AJ, Thomas J. Corticosteroids for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD003100. doi: 10.1002/14651858.CD003100.pub2. PMID 16625570